CLINICAL TRIAL: NCT00055315
Title: A Cognitive Group Treatment for Borderline Outpatients
Brief Title: Treatment for Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald Black, Professor of and MD in Psychiatry, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200112066; R01MH063746 (NIH); DATR A2-AIR
Record Dates: First submitted 2003-02-25; First posted 2003-02-26 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEPPS (Active Comparator): Patients with Borderline Personality Disorder. Each subject met DSM-IV criteria for BPD, confirmed through a clinical interview and a review of the patient's case notes
  Interventions: Behavioral: Systems Training for Emotional Predictability and Problem Solving (STEPPS)
- Treatment as Usual (Placebo Comparator): Patients with Borderline Personality Disorder. Each subject met DSM-IV criteria for BPD, confirmed through a clinical interview and a review of the patient's case notes.
  TAU for this BPD population includes medical management, group and individual therapy.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Systems Training for Emotional Predictability and Problem Solving (STEPPS) — STEPPS is a 20-week, manual-based, psychoeducational group treatment that combines skills training with cognitive-behavioral techniques. It includes a systems component to train family members, friends, and significant others.
  Arms: STEPPS
Behavioral: Treatment As Usual (TAU)
  Arms: Treatment as Usual

SUMMARY:
This study will expose patients to either a Systems Training for Emotional Predictability and Problem Solving (STEPPS) or treatment as usual (TAU) to determine the more effective therapy for treating borderline personality disorder.

DETAILED DESCRIPTION:
Participants are randomly assigned to receive either Systems Training for Emotional Predictability and Problem Solving (STEPPS) or treatment as usual (TAU) for 20 weeks. STEPPS is a new cognitive behavioral treatment which involves skills training for emotion management and lifestyle behaviors as well as education for the affected individual's family members, friends, and professional caregivers. Participants are assessed at baseline and Weeks 4, 8, 12, 16, and 20. Interviews of patient's health care providers and family members and self-rating scales are used to assess patients. Follow-up assessments are made 1, 3, 6, 9, and 12 months after study completion. Participants must live within a reasonable driving distance of Iowa City, IA.

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2002-07; Primary Completion 2007-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Roy J. and Lucille A. Carver College of Medicine, University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Blum N, Pfohl B, John DS, Monahan P, Black DW. STEPPS: a cognitive-behavioral systems-based group treatment for outpatients with borderline personality disorder--a preliminary report. Compr Psychiatry. 2002 Jul-Aug;43(4):301-10. doi: 10.1053/comp.2002.33497. PMID 12107867
- [Background] Black, D.W., Blum, N., Pfohl, B., & St. John, D: The STEPPS Group Treatment Program for Outpatients with Borderline Personality Disorder. Journal of Contemporary Psychotherapy 34:193-210, 2004.
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793